CLINICAL TRIAL: NCT01407913
Title: Efficacy Study of Caudal Epidural Steroid Injections in Patients With Low Back Pain/Radiculopathy
Brief Title: Caudal Epidural Steroid Injections for Low Back Pain/Sciatic Lumbar Pain
Acronym: FIA1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Assistant Professor of PMR, Orthopaedic Spine Surgeon, University of Ioannina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191/2010
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Pain; Disability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: caudal epidural steroid injection — injecting steroids in the epidural space via caudal route

SUMMARY:
The study hypothesis is that caudal epidural steroid injections provides short term relief to patients with persistent low back pain and sciatica due degenerative disc disease or lumbar spinal stenosis. Patients will be evaluated wiht clinical examination and radiological examinations before injections. They will be followed up with questionnaires on pain and disability up to 6 months postinjection.

ELIGIBILITY:
Inclusion Criteria:

* low back pain and sciatica due to lumbar disc herniation or lumbar spinals stenosis

Exclusion Criteria:

* infection, cancer, allergy to steroids or anesthetic, non controlled diabetes or hypertension, clotting disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
change from preinjection of oswestry disability index at 15 days and at 3-6 months postinjection | pre injection to 3-6 months postinjection
change from preinjection of Visual Analogue Scale at 15 days and at 3-6 months postinjection | preinjection to 3-6 months postinjection

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece